CLINICAL TRIAL: NCT04136808
Title: A Multicenter, Open-label, Expanded Access Treatment Protocol of Enfortumab Vedotin in Subjects With Locally Advanced or Metastatic Urothelial Carcinoma (EV-901)
Brief Title: An Expanded Access Treatment Protocol of Enfortumab Vedotin in Subjects With Locally Advanced or Metastatic Urothelial Carcinoma
Status: Approved for marketing | Type: Expanded Access
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 7465-CL-0108
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Locally Advanced or Metastatic Urothelial Carcinoma (UC)
Keywords: Locally Advanced or Metastatic Urothelial Carcinoma; enfortumab vedotin (EV); ASG-22CE; Expanded Access; EV-901
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — enfortumab vedotin

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: enfortumab vedotin (EV) — Participants will receive an intravenously (IV) administered dose once weekly for the first 3 weeks of every 4-week cycle (i.e., on days 1, 8, and 15)
  Other Names: ASG-22CE

SUMMARY:
The primary purpose of this expanded access program is to evaluate safety and tolerability of enfortumab vedotin (EV) in participants in the United States with locally advanced or metastatic urothelial carcinoma (UC) who have exhausted standard of care therapies and are not eligible to participate in an ongoing EV clinical study. This program will also evaluate the efficacy of EV.

DETAILED DESCRIPTION:
This treatment protocol is being conducted while a phase 3 enfortumab vedotin (EV) study is ongoing for participants with previously treated locally advanced or metastatic urothelial carcinoma (UC).

This is an expanded access program to provide EV to participants with locally advanced or metastatic UC who have previously been treated with a programmed cell death protein 1 (PD-1) or programmed death-ligand 1 (PD-L1) inhibitor, and a platinum containing regimen and for whom, in the judgment of the investigator, there is no available standard of care therapy. The participants must not be eligible for an ongoing EV clinical study. Participants who have previously participated in any EV studies or studies that included EV as one of the treatment options are not eligible, even if the participants was not given or assigned EV. To request enrollment, the investigator or designee will submit the candidate participant's relevant medical history and other records in order to support the participant's protocol eligibility.

Safety of EV will be assessed through evaluation of adverse events (AEs), serious adverse events (SAEs), Eastern Cooperative Oncology Group (ECOG) performance status, laboratory measurements, vital signs and physical examinations.

Participants will be provided with study medication until FDA approval and commercial availability of enfortumab vedotin (EV) or termination by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Subject has locally advanced or metastatic urothelial carcinoma (UC) and has progressed during or after the most recent therapy.
* Subject has previously received a platinum containing regimen (i.e., cisplatin or carboplatin) in the metastatic/locally advanced or neoadjuvant/adjuvant setting.

  * If the platinum containing regimen was administered in the adjuvant/neoadjuvant setting, progression on or after this treatment must be ≤ 12 months after treatment completion.
* Subject has previously received treatment with a programmed cell death protein 1 (PD-1) inhibitor or programmed death-ligand 1 (PD-L1) inhibitor (including, but not limited to, atezolizumab, pembrolizumab, durvalumab, avelumab and nivolumab) in the metastatic/locally advanced setting.

  * Subject treated with a PD-1 or PD-L1 inhibitor in the neoadjuvant/adjuvant setting and had recurrent or progressive disease either during therapy or ≤ 3 months of therapy completion may be enrolled.
* Subject has exhausted available standard of care therapies for locally advanced or metastatic UC.

  * Subject may have had any number of prior lines of therapy for locally advanced or metastatic UC.
* Subject has the following baseline laboratory data:

  * absolute neutrophil count ≥ 1500/mm3
  * platelet count ≥ 75 x 109/L
  * hemoglobin ≥ 8 g/dL
  * serum bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 3 x ULN for subjects with Gilbert's disease
  * creatinine clearance (CrCl) ≥ 15 mL/min or ≥ 30 mL/min for subjects with Eastern Cooperative Oncology Group (ECOG) performance status of 2 as estimated per institutional standards or as measured by 24 hour urine collection (glomerular filtration rate can also be used instead of CrCl)
  * alanine aminotransferase and aspartate aminotransferase ≤ 2.5 x ULN or ≤ 3 x ULN for subjects with liver metastases
* Subject has ECOG performance status of 0, 1 or 2.
* Female subject is not pregnant and at least 1of the following conditions apply:

  * not a woman of childbearing potential (WOCBP), or
  * a WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 6 months after final protocol treatment administration.
* Female subject must agree not to breastfeed starting at screening and throughout the treatment protocol period and for 6 months after final protocol treatment administration.
* Female subject must not donate ova starting at first dose of investigational product (IP) and throughout the treatment protocol period and for 6 months after final protocol treatment administration.
* Male subject with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 6 months after final protocol treatment administration.
* Male subject must not donate sperm during the treatment period and for 6 months after final protocol treatment administration.
* Male subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the treatment protocol period and for 6 months after final protocol treatment administration.
* Subject agrees not to participate in another interventional study while receiving treatment in the present treatment protocol.

Exclusion Criteria:

* Subject has ongoing sensory or motor neuropathy grade ≥ 2.
* Subject has ongoing clinically significant toxicity (grade 2 or higher with the exception of alopecia) associated with prior treatment (including systemic therapy, radiotherapy or surgery). Subject with hypothyroidism or panhypopituitarism related to treatment with PD-1 and PD-L1 inhibitors may be enrolled. Subject on hormone replacement therapy may be enrolled if on a stable dose.
* Subject has ongoing immunotherapy related myocarditis, colitis, uveitis or pneumonitis or other immunotherapy related toxicities requiring high doses of steroids (> 20 mg/day of prednisone or equivalent).
* Subject has previously received EV or enrolled in an EV study or a study that included EV as one of the treatment options (even if the subject was not given EV).
* Subject is a candidate for any ongoing EV clinical studies.
* Subject has known hypersensitivity to EV or to any excipient contained in the drug formulation of EV.
* Subject completed radiotherapy, major surgery or prior anticancer therapy ≤ 2 weeks before first EV dose.
* Subject has history of uncontrolled diabetes mellitus ≤ 3 months of the first EV dose. Uncontrolled diabetes is defined as hemoglobin A1C (HbA1c) ≥ 8% or HbA1c between 7 and < 8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
* Subject is currently receiving systemic antimicrobial treatment for viral, bacterial or fungal infection at the time of first dose of EV. Routine antimicrobial prophylaxis is permitted.
* Subject has recent history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction or cardiac symptoms (including congestive heart failure) consistent with New York Heart Association Classes III to IV that is not adequately treated and/or controlled at the time of first EV dose.
* Subject has other underlying medical condition that would impair the ability of the subject to receive or tolerate EV.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (15):
- United States (15):
  - UCLA Hematology Oncology, Los Angeles, California
  - John Wayne Cancer Institute, Santa Monica, California
  - St. Joseph Heritage Medical Group, Santa Rosa, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Community Hospital Anderson, Anderson, Indiana
  - New England Cancer Specialists, Topsham, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - NYU Langone Health, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - Inova Schar Cancer Institute, Fairfax, Virginia